CLINICAL TRIAL: NCT01236365
Title: Statins in Children With Type 1 Diabetes: Effects on Metabolism, Inflammation and Endothelial Function
Brief Title: Statins in Children With Type 1 Diabetes and Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Pfizer (Industry); Medtronic (Industry); Quest Diagnostics-Nichols Insitute (Industry)
Responsible Party: Principal Investigator, Nelly Mauras, Chief, Division of Endocrinology, Diabetes & Metabolism, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB# 185500
Record Dates: First submitted 2010-11-02; First posted 2010-11-08 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Insulin-Dependent; Hypercholesterolemia
Keywords: Type 1 diabetes; Children; Statins; Hypercholesterolemia; Lipoproteins; C reactive protein; Continuous glucose monitors; Adolescence; Abdominal magnetic resonance imaging; Toll like receptors; Receptors of advanced glycation end products; Nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Atorvastatin Placebo

INTERVENTIONS:
Drug: Atorvastatin — 10 or 20 mg daily
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Atorvastatin Placebo — 10 or 20 mg daily
  Arms: Placebo

SUMMARY:
Children with type1 diabetes (T1DM) have increased risk for cardiovascular disease (CVD) due to chronic increase in the blood sugars and inflammation. If there is also increased in cholesterol, it creates a highly abnormal environment not fully corrected by improved control of the blood sugars. CVD remains the principal risk of mortality in T1DM, and its prevention and treatment, compelling in children. This grant proposal encompasses 3 separate, yet interrelated projects addressing different aspects of CVD risk in children with T1DM. Project #1: a randomized controlled trial on the safety and efficacy of a class of drugs called "statins", which lower bad cholesterol in the body, in children with diabetes and elevated bad cholesterol. We will measure changes in concentration of blood inflammatory markers and for the 1st time, correlate levels of these markers with changes in blood sugar as measured by continuous glucose sensors, instruments that measure the blood sugar continuously through a small needle under the skin. Project #2: is a laboratory study to investigate the genetics and concentration of key molecules that participate in the inflammatory cascade and atheromatous plaque formation that causes CVD. Expression levels in children with T1DM will be compared with those in healthy controls for the 1st time. Project #3: examines the use of abdominal aortic MRI to measure damage to the arteries in children with T1DM and healthy age-matched controls. The results of these studies will likely provide important new data on the use of statins in children with diabetes.

ELIGIBILITY:
Inclusion Criteria:Project 1

* T1DM diagnosed clinically for > 1 year
* any HbA1C
* on stable insulin therapy
* Ages: 10 - 20 years
* both genders
* BMI < 85th percentile
* Fasting LDL-C>100mg/dl
* Normal thyroid function

Inclusion Criteria:Projects 2 and 3

* T1DM diagnosed clinically for > 3 year
* HbA1C > 8%
* on stable insulin therapy
* Ages: 12- 20 years
* both genders
* BMI < 85th percentile
* Fasting LDL-C>100mg/dl
* Normal thyroid function

Exclusion Criteria:Projects 1,2 and 3

* Severe dyslipidemia (LDL-C >160, TG > 400 mg/dl)
* Smoking
* Pregnancy
* Current use of anti-inflammatory or immunomodulatory drugs, lipid lowering, antidiabetic drugs
* Patients with hypertension and/or microalbuminuria will be allowed using balanced randomization and standardized treatment

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic 807 Children's Way Jacksonville, Florida 32207
Locations (5):
- United States (5):
  - Alfred I duPont Hospital, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Nemours Children's Clinic, Pensacola, Florida
  - Nemours Children's Clinic-Jefferson, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Canas JA, Ross JL, Taboada MV, Sikes KM, Damaso LC, Hossain J, Caulfield MP, Gidding SS, Mauras N. A randomized, double blind, placebo-controlled pilot trial of the safety and efficacy of atorvastatin in children with elevated low-density lipoprotein cholesterol (LDL-C) and type 1 diabetes. Pediatr Diabetes. 2015 Mar;16(2):79-89. doi: 10.1111/pedi.12245. Epub 2014 Nov 22. PMID 25418907
- [Result] McCulloch MA, Mauras N, Canas JA, Hossain J, Sikes KM, Damaso LC, Redheuil A, Ross JL, Gidding SS. Magnetic resonance imaging measures of decreased aortic strain and distensibility are proportionate to insulin resistance in adolescents with type 1 diabetes mellitus. Pediatr Diabetes. 2015 Mar;16(2):90-7. doi: 10.1111/pedi.12241. Epub 2014 Dec 18. PMID 25524487

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: 10 or 20 mg daily
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 21 | 21
Completed | 19 | 19
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Moved Out of State | 1 | 0
Not completed — Dropped at Randomization due to high LFT | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (2.2) | 15.4 (2.7) | 15.1 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  non-Hispanic white | 17 | 14 | 31
  Other | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: LDL-C Levels Assessed at Randomization and 6 Months
Description: To assess if the use of statins in children with type 1 DM is safe, improves measures of LDL-C. Subjects will have a physical exam, laboratories, nutritional counseling and moderate aerobic exercise recommended. Diabetes management will be intensified. At 3 months fasting lipoprotein fractions (ion mobility)re-drawn and if LDL-C >100mg/dl patients will be randomized to treatment with statins or placebo for 6 months, randomization stratified by BP and microalbuminuria, duration of diabetes and HgA1C. At 1 month safety labs will be repeated and blood withdrawn again at 3 and 6 months from baseline.
Time Frame: Randomization and 6 months
Population: Project #1. Adjusted for age, gender and ISS (Insulin sensitivity score)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Atorvastatin LDL-C at Randomization | Atorvastatin LDL-C at 6 Months | Placebo LDL-C at Randomization | Placebo LDL-C at 6 Months
Number analyzed (Participants) | 19 | 19 | 19 | 19
mg/dL | 128 (4) | 87 (5) | 126 (5) | 133 (8)
Statistical Analysis 1: Comparison: Atorvastatin LDL-C at Randomization vs Atorvastatin LDL-C at 6 Months; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Change in LDL-C between Atorvastatin and Placebo

2. Primary Outcome: Hs-CRP Levels Assessed at Randomization and 6 Months
Description: To assess if the use of statins in children with type 1 DM decreases the concentration of inflammatory markers.
Time Frame: Randomization and 6 months
Population: Project #1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Atorvastatin hsCRP at Randomization | Atorvastatin hsCRP at 6 Months | Placebo hsCRP at Randomization | Placebo hsCRP at 6 Months
Number analyzed (Participants) | 19 | 19 | 19 | 19
mg/dL | 0.363 [0.148 to 0.817] | 0.419 [0.165 to 1.092] | 0.248 [0.149 to 0.959] | 0.446 [0.181 to 0.958]
Statistical Analysis 1: Comparison: Atorvastatin hsCRP at Randomization vs Atorvastatin hsCRP at 6 Months vs Placebo hsCRP at Randomization vs Placebo hsCRP at 6 Months; Test type: Superiority or Other; p = 0.913, Wilcoxon (Mann-Whitney) — Change in hsCRP (6months minus 0months) between Atorvastatin and Placebo

3. Secondary Outcome: MAGE
Description: Mean amplitude of glycemic excursion (MAGE) with continuous glucose monitoring (CGM - IPro®, Medtronic Minimed) worn blindly for 6d to assess glucose variability
Time Frame: Randomization and 6 months
Population: Project #1. 4 Atorvastatin and 8 Placebo Subjects did not complete their CGM at 6months.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Atorvastatin MAGE at Randomization | Atorvastatin MAGE at 6 Months | Placebo MAGE at Randomization | Placebo MAGE at 6 Months
Number analyzed (Participants) | 19 | 15 | 19 | 11
mg/dL | 150 (9) | 156 (13) | 156 (6) | 152 (8)

4. Secondary Outcome: RAGE
Description: Receptor for Advanced Glycation End Products
Time Frame: Randomization and 6 months
Population: Project #2. Study Subjects were given the option to participate in the Project #2 genetic substudy; 9 Atorvastatin and 12 Placebo Subjects participated in Project #2. 1 Atorvastatin and 1 Placebo Subject did not complete the 6 month genetic test.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Atorvastatin LDL-C at Randomization | Atorvastatin LDL-C at 6 Months | Placebo LDL-C at Randomization | Placebo LDL-C at 6 Months
Number analyzed (Participants) | 9 | 8 | 12 | 11
pg/mL | 49 (11) | 35 (5) | 50 (7) | 58 (17)

5. Secondary Outcome: Descending Aortic Strain
Description: Subclinical atherosclerosis and arterial stiffness of abdominal aortic MRI
Time Frame: Randomization
Population: Project #3. Study Subjects were given the option to participate in the Project #3 MRI substudy; 11 Atorvastatin and 8 Placebo Subjects participated in Project #3.
Measure: Mean (Standard Deviation); unit: percent area change
Arm/Group | Atorvastatin at Randomization | Placebo at Randomization
Number analyzed (Participants) | 11 | 8
percent area change | 27.2 (6.4) | 29 (8.5)
Statistical Analysis 1: Comparison: Atorvastatin at Randomization; Test type: Other; p = 0.09, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21
Other Adverse Events (participants affected / at risk) | 11/21 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=21) | Placebo (N=21)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fell from horse and sustained a concussion and fractured finger
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=21) | Placebo (N=21)
Cut/Laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Stomach Discomfort (Gastrointestinal disorders) | 2 (2) | 3 (3)
Acid Reflux (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hematuria with Flank Pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lower Extremity Cramping (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Hand Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinus Symptoms (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Throat Infection (Infections and infestations) | 2 (2) | 1 (3)
Abnormal Chemistry Labs (Hepatobiliary disorders) | 1 (1) | 1 (2)
Elevated CK Blood Level (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hypoglycemic Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (Social circumstances) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes